CLINICAL TRIAL: NCT00770133
Title: A Multi-center, Double-masked, Randomized, Placebo-controlled Evaluation of the Onset and Duration of Action of KetoNaph Ophthalmic Solution in the Conjunctival Allergen Challenge (CAC) Model of Acute Allergic Conjunctivitis.
Brief Title: Ketotifen/Naphazoline Ophthalmic Solution in the Conjunctival Allergen Challenge Model of Acute Allergic Conjunctivitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 572
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Ketotifen; Naphazoline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ketotifen/naphazoline (Experimental): Ketotifen/naphazoline ophthalmic solution administered in either the right eye, left eye or both eyes at visit 3 and visit 4.
  Interventions: Drug: Ketotifen/naphazoline
- Vehicle (Placebo Comparator): Vehicle of ketotifen/naphazoline ophthalmic solution administered in either the right eye, left eye or both eyes at visit 3 and visit 4.
  Interventions: Drug: Vehicle
- Naphazoline (Active Comparator): Naphazoline ophthalmic solution administered in either the right eye, left eye or both eyes at visit 3 and visit 4.
  Interventions: Drug: Naphazoline
- Ketotifen (Active Comparator): Ketotifen ophthalmic solution administered in either the right eye, left eye or both eyes at visit 3 and visit 4.
  Interventions: Drug: Ketotifen

INTERVENTIONS:
Drug: Ketotifen/naphazoline — One drop of ketotifen fumarate 0.025% and naphazoline HCl 0.05% ophthalmic solution at visit 3 and visit 4.
  Arms: Ketotifen/naphazoline
Drug: Naphazoline — One drop of naphazoline HCl 0.05% ophthalmic solution at visits 3 and 4.
  Arms: Naphazoline
Drug: Ketotifen — One drop of ketotifen fumarate 0.025% ophthalmic solution at visits 3 and 4.
  Arms: Ketotifen
Drug: Vehicle — One drop of vehicle ophthalmic solution at visit 3 and visit 4.
  Arms: Vehicle

SUMMARY:
The purpose of this study is to establish the safety and efficacy of ketotifen/naphazoline ophthalmic solution compared to vehicle and its individual components in alleviating the signs and symptoms of conjunctival allergen challenge (CAC)-induced allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Positive history of ocular allergies and positive skin test reaction to cat hair, cat dander, grasses, ragweed, and/or trees within the past 24 months.
* Calculated best-corrected visual acuity of 0.7 logMAR or better in each eye as measured using the ETDRS chart.
* Positive bilateral conjunctival allergen challenge(CAC) reaction within 10 minutes of instillation of the last titration of allergen at visit 1.
* Positive bilateral CAC reaction for at least 2 out of 3 time points at visit 2.

Exclusion Criteria:

* Known contraindications or sensitivities to the study medication or its components.
* Any ocular condition that, in the opinion of the investigator, could affect the subjects safety or trial parameters.
* Use of disallowed medications during the period indicated prior to study enrollment or during the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Trusso, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Ophthalmic Research Consultants, Inc., North Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 70 eyes in the KetoNaph group, 72 in the ketotifen group, 70 in the naphazoline group, and 70 in the vehicle group, for a total of 282 eyes (141 subjects).
Period: Overall Study
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle
Started | 35 | 36 | 35 | 35
Completed | 32 | 35 | 32 | 32
Not Completed | 3 | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle | Total
Number analyzed (Participants) | 35 | 36 | 35 | 35 | 141
Age, Continuous [Mean (Full Range); unit: years] | 36.1 [15 to 71] | 40.7 [15 to 71] | 38.2 [16 to 76] | 38.4 [16 to 76] | 38.4 [15 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 18 | 18 | 73
  Male | 19 | 15 | 17 | 17 | 68

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Ocular itching was evaluated by the participant at 3, 5, and 7 minutes post challenge. Assessments were made using a 0-4 numerical analog scale, allowing 0.5-unit increments (but disallowing 0.25-unit increments), where: 0.0=None and 4.0=Incapacitating itch with an irresistible urge to rub
Time Frame: 3, 5, and 7 minutes post challenge at 14 days
Population: The intent to treat population consisted of participants who were randomized, received investigational treatment, and had at least 1 post-challeng assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 34 | 36 | 34 | 35
Number analyzed (eyes) | 68 | 72 | 68 | 70
score on a scale
  3 minutes post-challenge | 0.43 (0.62) | 0.40 (0.65) | 1.60 (0.92) | 1.81 (0.88)
  5 minutes post-challenge | 0.65 (0.76) | 0.59 (0.79) | 1.67 (1.01) | 1.96 (0.94)
  7 minutes post-challenge | 0.60 (0.83) | 0.56 (0.87) | 1.54 (0.96) | 1.84 (1.01)

2. Primary Outcome: Conjunctival Redness
Description: Conjunctival hyperemia was evaluated by the Investigator at 7, 15, and 20 minutes post challenge. Assessments were completed using a 0-4 numerical analog scale, allowing 0.5-unit increments, where: 0.0=None and 4.0=Extremely severe.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 34 | 36 | 34 | 35
Number analyzed (eyes) | 68 | 72 | 68 | 70
score on a scale
  7 minutes post-challeng | 0.89 (0.87) | 1.49 (0.83) | 1.63 (0.84) | 2.06 (0.77)
  15 minutes post-challenge | 1.13 (1.00) | 1.80 (0.87) | 1.69 (0.89) | 2.26 (0.78)
  20 minutes post-challenge | 1.13 (1.02) | 1.88 (0.89) | 1.57 (0.92) | 2.18 (0.85)

3. Secondary Outcome: Ciliary Redness
Description: Ciliary hyperemia (redness) was evaluated by the Investigator at 7, 15, and 20 minutes post challenge. Assessments were made using the same 0-4 scale, allowing 0.5-unit increments, where: 0.0=None and 4.0=Extremely severe.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: This outcome measure was not assessed for the Vehicle group. The intent to treat population consisted of participants who were randomized, received investigational treatment, and had at least 1 post-challenge assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 34 | 36 | 34 | 0
Number analyzed (eyes) | 68 | 72 | 68 | 0
score on a scale
  7 minutes post-challenge | 0.81 (0.86) | 1.33 (0.88) | 1.49 (0.89) |
  15 minutes post-challenge | 1.05 (1.05) | 1.76 (0.91) | 1.59 (0.91) |
  20 minutes post-challenge | 1.04 (1.03) | 1.76 (0.94) | 1.54 (0.92) |

4. Secondary Outcome: Episcleral Redness
Description: Episcleral hyperemia (redness) was evaluated by the Investigator at 7, 15, and 20 minutes post challenge. Assessments were made using the same 0-4 scale, allowing 0.5-unit increments, where: 0.0=None and 4.0=Extremely severe.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 34 | 36 | 34 | 0
Number analyzed (eyes) | 68 | 72 | 68 | 0
score on a scale
  7 minutes post-challenge | 0.91 (0.89) | 1.51 (0.85) | 1.65 (0.86) |
  15 minutes post-challenge | 1.17 (1.01) | 1.76 (0.88) | 1.68 (0.94) |
  20 minutes post-challenge | 1.15 (1.03) | 1.88 (0.90) | 1.60 (0.94) |

5. Secondary Outcome: Chemosis
Description: Chemosis was evaluated by the Investigator at 7, 15, and 20 minutes post challenge on a 0-4 numerical analog scale, allowing 0.5-unit increments, where: 0.0=None and 4.0=Extremely severe.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 34 | 36 | 34 | 0
Number analyzed (eyes) | 68 | 72 | 68 | 0
score on a scale
  7 minutes post-challenge | 0.27 (0.33) | 0.28 (0.30) | 0.39 (0.40) |
  15 minutes post-challenge | 0.34 (0.38) | 0.46 (0.47) | 0.54 (0.55) |
  20 minutes post-challenge | 0.39 (0.41) | 0.49 (0.46) | 0.54 (0.58) |

6. Secondary Outcome: Eyelid Swelling
Description: Lid swelling was evaluated by the participant at 7, 15, and 20 minutes post challenge on a 0-3 numerical analog scale, with 0.5-unit increments disallowed, where: 0.0=None and 3.0=Severe.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 34 | 36 | 34 | 0
Number analyzed (eyes) | 68 | 72 | 68 | 0
score on a scale
  7 minutes post-challenge | 0.2 (0.4) | 0.2 (0.4) | 0.2 (0.4) |
  15 minutes post-challenge | 0.2 (0.5) | 0.2 (0.4) | 0.2 (0.4) |
  20 minutes post-challenge | 0.2 (0.5) | 0.2 (0.4) | 0.2 (0.4) |

7. Secondary Outcome: Percentage of Eyes With hTearing
Description: Tearing was evaluated by the participant at 7, 15, and 20 minutes post challenge. Tearing was recorded as either absent or present.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: as for outcome 3
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 34 | 36 | 34 | 0
Number analyzed (eyes) | 68 | 72 | 68 | 0
eyes
  7 minutes post-challenge | 7 | 11 | 13 |
  15 minutes post-challenge | 4 | 9 | 12 |
  20 minutes post-challenge | 5 | 6 | 11 |

8. Secondary Outcome: Percentage of Eyes With Ocular Mucus Discharge
Description: Ocular mucous discharge was evaluated by the Investigator at 7, 15, and 20 minutes post challenge. Mucous discharged was recorded as either absent or present.
Time Frame: 7, 15, and 20 minutes post challenge at 14 days
Population: as for outcome 3
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle
Number analyzed (Participants) | 34 | 36 | 34 | 0
Number analyzed (eyes) | 68 | 72 | 68 | 0
eyes
  7 minutes post-challenge | 0 | 0 | 0 |
  15 minutes post-challenge | 0 | 0 | 0 |
  20 minutes post-challenge | 0 | 0 | 0 |

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Ketotifen/Naphazoline | Ketotifen | Naphazoline | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.